CLINICAL TRIAL: NCT05410405
Title: Changes in Implant Stability Using Different Site Preparation Techniques: Osseodensification Drills Versus Piezoelectric Surgery. A Multicenter Randomized Controlled Clinical Trial
Brief Title: Osseodensification Drills Versus Piezoelectric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Foggia (Other); University of Trieste (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: piezodensi
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Investigator
Masking Description: implant stability assessment was blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 millimeter implants (Experimental): implant insertion with piezo surgical osteotomy and with osseodensification drills
  Interventions: Procedure: implant site preparation
- 10 millimeter implants (Experimental): implant insertion with piezo surgical osteotomy and with osseodensification drills
  Interventions: Procedure: implant site preparation

INTERVENTIONS:
Procedure: implant site preparation — piezoelectric bone surgery osseodensification drills
  Other Names: implant insertion

SUMMARY:
implant stability is the first requirement for implant success. the aim is to assess whether different implant site preparation technique may impact the value of the primary stability.

DETAILED DESCRIPTION:
Impianti stability represents one of the most fundamental issue for implant success. Different techniques of implant site preparation are available such as twist drill, osteotome, piezosurgery and lastly, osseodensification. Due to their different approach an biological rationale, piezosurgery and osseodensification might show diverse impact on implant first and secondary stability, therefore the aim of the present study was the assessment of primary and secondary stability changes of values between implant sites prepared with piezoelectric bone surgery and with specific osseodensification drills.

Patients with bilateral single maxillary edentulism will randomly receive implant site preparation with piezoelectric approach or with osseodensification drills. standardized implants will be therefore inserted and primary stability will be assessed at the time of implant insertion and during the subsequent timepoints.

ELIGIBILITY:
Inclusion Criteria:

* bilateral single maxillary edentulism

Exclusion Criteria:

* smoking habit
* history of periodontal disease
* uncontrolled diabetes
* pregnancy or breastfeeding
* head and neck radiotherapy or chemotherapy
* bone antiresorptive therapy
* coagulopaties

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
implant insertion torque | at implant insertion
  insertion torque
implant stability quotient | at implant insertion
  resonance frequency

SECONDARY OUTCOMES:
implant secondary stability | 7 days after implant insertion
  resonance frequency
implant secondary stability | 14 days after implant insertion
  resonance frequency
implant secondary stability | 21 days after implant insertion
  resonance frequency
implant secondary stability | 28 days after implant insertion
  resonance frequency
implant secondary stability | 2 months after implant insertion
  resonance frequency
implant secondary stability | 3 months after implant insertion
  resonance frequency

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Director — International Piezoelectric Surgery Academy
Locations (2):
- Italy (2):
  - Hesire, Cassano Allo Ionio, CS
  - Piezosurgery Academy, Parma

IPD SHARING:
Plan to Share IPD: No
no sharing is planned